CLINICAL TRIAL: NCT03013439
Title: Phase I Dose-escalation Trial of the Safety, Pharmacokinetics, and Pharmacodynamics of Iron Isomaltoside (Monofer®) Administered as Single Bolus Injections or Infusions in Japanese Subjects With Iron Deficiency Anemia
Brief Title: Dose-escalation Trial of the Safety, Pharmacokinetics, and Pharmacodynamics of Iron Isomaltoside (Monofer®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PK-IDA-01
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-01

CONDITIONS: Anemia; Deficiency Diseases; Anemia, Iron Deficiency; Hematologic Disease; Iron Metabolism Disorders
MeSH Terms: conditions — Anemia; Deficiency Diseases; Anemia, Iron-Deficiency; Hematologic Diseases; Iron Metabolism Disorders | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- cohort 1 iron isomaltoside (Experimental): treated with first dose level of iron isomaltoside
  Interventions: Drug: Iron Isomaltoside
- cohort 2 iron isomaltoside (Experimental): treated with second dose level of iron isomaltoside
  Interventions: Drug: Iron Isomaltoside
- cohort 3 iron isomaltoside (Experimental): treated with third dose level of iron isomaltoside
  Interventions: Drug: Iron Isomaltoside
- cohort 4 iron isomaltoside (Experimental): treated with fourth dose level of iron isomaltoside
  Interventions: Drug: Iron Isomaltoside

INTERVENTIONS:
Drug: Iron Isomaltoside — The trial is a dose escalating trial.
  Other Names: Monofer

SUMMARY:
The trial is an open-label, 4 cohorts, sequential, dose-escalating, single dose trial.

DETAILED DESCRIPTION:
IDA is highly prevalent in subjects with cancer and gastrointestinal diseases such as inflammatory bowel diseases, menstruating or pregnant women, and subjects who have undergone bariatric procedure. IDA can have a substantial medical and quality of life (QoL) burden on the subjects, and treatment of these subjects includes controlling the bleeding and replenishing lost iron.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese man or woman ≥ 20 years, < 65 years of age
2. Hb of ≥ 9.0 g/dL, < 12.0 g/dL for women and < 13.0 g/dL for men
3. Serum ferritin < 25 ng/mL
4. TIBC ≥ 360 μg/dL
5. Body weight ≥ 50 kg
6. Willingness to participate and signing the informed consent form

Exclusion criteria include:

1. Anemia caused by conditions other than iron deficiency
2. Cancer
3. IV or oral iron treatment, or blood transfusion 4 weeks prior to screening
4. Erythropoiesis stimulating agent (ESA) treatment prior to screening
5. Imminent expectation of blood transfusion on part of treating physician
6. Iron overload or disturbances (e.g. hemochromatosis and hemo-siderosis)
7. Known hypersensitivity reaction to iv iron preparations
8. Decompensated liver cirrhosis or active hepatitis
9. Active acute or chronic infections
10. Pregnant or nursing women.
11. Planned elective surgery during the trial

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-06-04 (Actual)

PRIMARY OUTCOMES:
Proportion of adverse events | 1 week
  Proportion of adverse events will be collected and evaluated for relatedness, severity, seriousness, and expectedness.

SECONDARY OUTCOMES:
Maximum plasma drug concentration [Cmax] | 1 week
Area Under the Curve [AUC] | 1 week
Time to reach one-half of the maximum drug concentration [T1/2] | 1 week
Time to reach maximum drug concentration [Tmax] | 1week
Change in concentration of hemoglobin (g/dL) | 1 week
Change in concentration of serum ferritin (ng/mL) | 1 week
Change in concentration of total iron binding capacity (μg/dL ) | 1 week
Change in concentrations of transferrin saturation (%) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Ikebukuro, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No